CLINICAL TRIAL: NCT06064383
Title: Epidemiology and Risk Factors of Suicidal Attacks in Children and Adolescents at Assiut University Children Hospital
Brief Title: Suicidal Attacks in Children and Adolescents
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Ramadan Abd El-Hafiz, Assistant lecturer, Assiut University
Other Study IDs: suicidal attacks in children
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Suicidal Attacks

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: suicide attacks — select the most common causes, risk factors, methods and circumstances surrounding suicidal attempts in children and adolescents at aaiut university children hospital

SUMMARY:
Discuss suicidal behaviors among children and adolescents at Assiut university children hospital (AUCH) and Select the most common causes, risk factors, methods and circumstances surrounding suicidal attempts in children and adolescents at AUCH. Also, Estimate incidence of children and adolescents with suicidal attempts at AUCH.

DETAILED DESCRIPTION:
Suicide is a major public health problem that affects people of all ages, including children and adolescents. A child's decision to commit suicide is influenced by many social and psychological factors, as well as mental illness and addiction. Suicide is defined as death caused by self-directed injurious behavior with an intent to die as a result of the behavior; suicide attempt is defined as a nonfatal, self-directed, potentially injurious behavior with an intent to die as a result of the behavior even if the behavior does not result in injury; and suicidal ideation is defined as thinking about, considering, or planning suicide.

Suicide is the fourth leading cause of death worldwide among 15-29 year-olds (WHO, 2021). Globally, lifetime prevalence rates are approximately 9.2% for suicidal ideation and 2.7% for suicide attempt.

The leading methods of suicide for the 15- to 19-year age group in 2013 were suffocation (43%), discharge of firearms (42%), poisoning (6%), and falling (3%). It is estimated that around 20% of global suicides are due to pesticide self-poisoning, most of which occur in rural agricultural areas in low- and middle-income countries. The availability of potentially lethal drugs may also increase the risk of suicide or at least increase the medical lethality of an attempt.

Although no specific tests are capable of identifying a suicidal person, specific risk factors exist. Some risk factors for suicide can be classified as being modifiable or non-modifiable. Modifiable risk factors are dynamic and may be influenced by treatment (eg. suicidal ideation, current stressors and poor physical health). Non-modifiable risk factors are static and do not change over time (eg. family history of suicide or suicide attempts, history of adoption, male gender, parental mental health problems, history of physical or sexual abuse, and a previous suicide attempt). Personal mental health problems that predispose to suicide include sleep disturbances, depression, substance use disorders, and pathologic Internet use. Social and environmental risk factors include bullying, impaired parent-child relationship, living outside of the home (homeless or in a corrections facility or group home), difficulties in school, social isolation, and presence of stressful life events. Youth seem to be at much greater risk from media exposure than adults and may imitate suicidal behavior seen on television. Media coverage of an adolescent's suicide may lead to cluster suicides, with the magnitude of additional deaths proportional to the amount, duration, and prominence of the media coverage.

The first step in treating a child after a suicide attempt is a control of the vital signs of the patient. The priority is to reverse the life-threatening condition, and then to treat the disease . Options for immediate evaluation include hospitalization, transfer to an emergency department, or a same-day appointment with a mental health professional. Adolescents with a responsive and supportive family, little likelihood of acting on suicidal impulses (e.g., thought of dying with no intent or plan for suicide), and someone who can take action if there is mood or behavior deterioration may require only outpatient treatment.

ELIGIBILITY:
Inclusion Criteria:

* All children between the ages of 5-18 years, with at least history of one suicidal attempt.

Exclusion Criteria:

* • Adult population and don't include children and adolescents as participants. Children and adolescents committing suicide by gunshots and falling from height.

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children between the ages of 5-18 years, with at least history of one suicidal attempt . Children and adolescents committing suicide by gunshots and falling from height not incuded.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Epidemiology and Risk factors of suicidal attacks in children and adolescents | 1 year
  Select the most common causes, risk factors, methods and circumstances surrounding suicidal attempts in children and adolescents.Also, Estimate Percentage of children and adolescents with suicidal attempts at assiut university children hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Khalaf Abd El-Aal Sayed, Dr, Study Director — Assiut University; Emad El-Deen Mohamoud, Dr, Principal Investigator — Assiut University

REFERENCES:
- [Background] Klonsky ED, May AM, Saffer BY. Suicide, Suicide Attempts, and Suicidal Ideation. Annu Rev Clin Psychol. 2016;12:307-30. doi: 10.1146/annurev-clinpsy-021815-093204. Epub 2016 Jan 11. PMID 26772209
- [Background] Berk MS. Editorial: Suicide prevention in youth. Child Adolesc Ment Health. 2022 Nov;27(4):325-327. doi: 10.1111/camh.12604. PMID 36250453
- [Background] Ike K, Haginoya K, Suzuki Y, Yokoyama H, Iinuma K, Numazaki Y, Soga T, Tada K. A case of chronic mumps virus encephalitis manifesting intractable epileptic seizures. Jpn J Psychiatry Neurol. 1990 Jun;44(2):356-7. No abstract available. PMID 2259024
- [Background] Bridge JA, Goldstein TR, Brent DA. Adolescent suicide and suicidal behavior. J Child Psychol Psychiatry. 2006 Mar-Apr;47(3-4):372-94. doi: 10.1111/j.1469-7610.2006.01615.x. PMID 16492264
- [Background] Gordon M, Melvin G. Risk assessment and initial management of suicidal adolescents. Aust Fam Physician. 2014 Jun;43(6):367-72. PMID 24897985
- [Background] Chun TH, Katz ER, Duffy SJ, Gerson RS. Challenges of managing pediatric mental health crises in the emergency department. Child Adolesc Psychiatr Clin N Am. 2015 Jan;24(1):21-40. doi: 10.1016/j.chc.2014.09.003. Epub 2014 Oct 3. PMID 25455574
- See also: WHO (World Health Organ.). 2014. Preventing suicide: a global imperative. — http://apps.who.int/iris/bitstream/10665/131056/1/9789241564779-eng.pdf?ua=1.